CLINICAL TRIAL: NCT01083797
Title: Sedation to Electroencephalography With Dexmedetomidine or Chloral Hydrate: a Comparative Study of the Qualitative and Quantitative Electroencephalogram Pattern
Brief Title: Sedation to Electroencephalography With Dexmedetomidine or Chloral Hydrate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Santa Casa de Misericórdia de Belo Horizonte (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, Magda Lourenço Fernandes, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 106/2009
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Other Conditions of Brain
Keywords: Sedation; Electroencephalography; Dexmedetomidine; Chloral hydrate
MeSH Terms: interventions — Dexmedetomidine; Chloral Hydrate; Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dexmedetomidine, chloral hydrate (Other): sedation with dexmedetomidine or chloral hydrate on separate occasions in the same patients
  Interventions: Drug: Dexmedetomidine; Drug: Chloral Hydrate

INTERVENTIONS:
Drug: Dexmedetomidine — 1 μg kg-1 infused in 10 min, and thereafter maintained from 0.2 to 0.7 μg kg-1 h- 1
  Other Names: Dexmedetomidine: Precedex, Abbott Laboratories
Drug: Chloral Hydrate — Initial dose=50 mg/kg
  Other Names: Chloral Hydrate 10% solution (100 mg/ml)

SUMMARY:
This study evaluates the use of dexmedetomidine or chloral hydrate for sedation during electroencephalography in patients with neurological disorders. The hypothesis is that this drugs provides similar changes in EEG pattern.

DETAILED DESCRIPTION:
Patients with chronic neurological disorders such as cerebral palsy or autism need to be sedated during electroencephalography (EEG). However, various sedatives and hypnotics affect the outcome of the review and is not shown. Chloral hydrate (CH) is widely used in children, but in this patients it is less effective.Recently, dexmedetomidine (DEX) has been tested because preliminary data suggests that this drug does not affect the EEG. The aim of the present work was to compare the electroencephalogram (EEG) pattern during CH or DEX sedation, to test the hypothesis that both drugs exert similar effects in EEG.Seventeen patients were evaluated during sedation with DEX or CH on separate occasions.The EEG was subjected to qualitative and quantitative analysis. Clinical variables were also compared.

ELIGIBILITY:
Inclusion Criteria:

* neurological disorder
* behavior disorder
* epilepsy

Exclusion Criteria:

* cardiac disease
* respiratory disease

Ages: 12 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
electroencephalogram pattern | twenty minutes
  Qualitative analysis: identification of the deepest phase of sleep achieved during the examination, evaluation of background activity (normal, fast activity increased or slow activity increased).
  Quantitative analysis: density, duration, and amplitude of sleep spindles, spectral power and dominant frequence.

SECONDARY OUTCOMES:
Effective sedative | twenty minutes
  Maintain adequate sedation permitting the completion of the examination
Adverse effects | Two hours
  Incidence of bradycardia, hypotension, respiratory complications and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Magda Fernandes, Principal Investigator — Santa Casa de Misericórdia de Belo Horizonte; Gomez Renato, Study Director — Federal University of Minas Gerais
Locations (1):
- Santa Casa de Belo Horizonte, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Lubisch N, Roskos R, Berkenbosch JW. Dexmedetomidine for procedural sedation in children with autism and other behavior disorders. Pediatr Neurol. 2009 Aug;41(2):88-94. doi: 10.1016/j.pediatrneurol.2009.02.006. PMID 19589455
- [Background] Huupponen E, Maksimow A, Lapinlampi P, Sarkela M, Saastamoinen A, Snapir A, Scheinin H, Scheinin M, Merilainen P, Himanen SL, Jaaskelainen S. Electroencephalogram spindle activity during dexmedetomidine sedation and physiological sleep. Acta Anaesthesiol Scand. 2008 Feb;52(2):289-94. doi: 10.1111/j.1399-6576.2007.01537.x. Epub 2007 Nov 14. PMID 18005372